CLINICAL TRIAL: NCT02084290
Title: Evaluating a Prediction Tool and Decision Aid for Patients With Crohn's Disease
Brief Title: Evaluating a Shared Decision Making Program for Crohn's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); University of Pittsburgh (Other); MOUNT SINAI HOSPITAL (Other); Cedars-Sinai Medical Center (Other); University of Maryland (Other); Brigham and Women's Hospital (Other); Thomas Jefferson University (Other); University of Chicago (Other); Atlanta Gastroenterology Associates (Other); Long Island Clinical Research Associates (Unknown); Center for Digestive and Liver Diseases (Unknown); Charlotte Gastroenterology and Hepatology (Unknown); Minnesota Gastroenterology (Unknown); Ohio Gi and Liver Institute (Unknown); Winthrop University Hospital (Other)
Responsible Party: Principal Investigator, Corey Siegel, Section Chief, Section of Gastroenterology, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AHRQR01 HS21747 D13129; R01HS021747 (AHRQ)
Record Dates: First submitted 2014-01-29; First posted 2014-03-11 (Estimated); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease; Shared Decision Making; Decision Aid
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Shared Decision Making Program (Experimental): Patients will have access to an educational decision making program and a risk prediction model, this web based program will be sent subjects in the intervention arm upon enrollment, they can access the program as many times as they wish.
  Interventions: Behavioral: Shared Decision Making Program
- Control (No Intervention): Subjects enrolled at sites participating as control arms will access the same web-based surveys as the intervention group, and receive the same contacts from the study coordinator as the subjects enrolled at intervention sites.

INTERVENTIONS:
Behavioral: Shared Decision Making Program — This study is cluster randomized by study-site, Subjects enrolled at intervention sites will access an educational program and risk prediction tool. Their decisions about treatments will be compared to subjects that did not view the educational program or risk prediction tool.
  Arms: Shared Decision Making Program

SUMMARY:
Specific Aim: Study the impact of the Crohn's Disease Shared Decision Making Program on patients' treatment choice, persistence with chosen therapy, decision quality, cost of care, and outcomes

Hypothesis: The Crohn's Disease Shared Decision Making Program will help patients understand which treatments are right for them and will lead to a higher acceptance of appropriate therapy, improved persistence with chosen therapy, lower costs and improved clinical outcomes. To accomplish this aim, Investigators will perform a randomized controlled trial to:

1. Determine how the shared decision making program influences patients' choice of therapy
2. Evaluate how the shared decision making program affects persistence with chosen therapy
3. Determine how the shared decision making program affects decision quality
4. Determine how the shared decision making program influences cost of care and clinical outcomes

Expected Outcome and Impact: Investigators expect that this program will influence patients' choice of therapy, persistence with their preferred therapy, and lead to improved clinical outcomes. Investigators believe that this product can be successfully operationalized in the clinic to establish a new paradigm of how providers can communicate personalized treatment options to patients across a broad range of diseases.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Crohn's Disease based on standard clinical, radiographic, endoscopic, and histologic criteria
* Age 18 or older
* Fluent, English Speaking
* A candidate to receive immunomodulators or anti-TNF therapy based on their providers recommendation
* not currently taking immunomodulators (6-mercapropurine, azathioprine, methotrexate) or anti-TNF agents (infliximab, adalimumab, certolizumab pegol)

Exclusion Criteria:

* Participant in a pilot study/focus group for development of Crohn's Shared Decision Making Program
* Currently taking any medication that is contraindicated to take together with an immunomodulator or anti-TNF agent
* Known intolerance to either immunomodulators or anti-TNF agents
* Lack of accessibility to e-mail for follow-up surveys

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2014-03; Primary Completion 2017-08-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion of patients choosing Combination therapy | Week 1

SECONDARY OUTCOMES:
Time to initiation of therapy | Week 1, Week 2, week 26, week 52, week 78, week 110
Patient Choice of therapy | Week 1, Week 2, week 26, week 52, week 78, week 110
  no therapy, immunomodulator monotherapy, anti-TNF monotherapy, Combination therapy
Persistence (adherence) with chosen therapy | Week 1, Week 2, week 26, week 52, week 78, week 110
Quality of Decision | Week 1, Week 2, week 26, week 52, week 78, week 110
  i. Decisional conflict (validated scale) ii. Decision consistent with patient values (i.e., patient receiving the treatment that they want) iii. Trust in physician
Cost of Care | week 110
  Crohn's disease related costs at 2 years
Remission | 6 months, 1 year, 2 years
  Proportion of patients in clinical remission
Patients on Steroids | 6 months, 1 year, 2 years
  Proportion of patients taking steroids
Surgeries | 6 months, 1 year, 2 years
  Proportion of patients requiring Crohn's disease related surgery
Crohn's disease related hospitalizations | 6 months, 1 year, 2 years
  Number of hospitalizations

CONTACTS AND LOCATIONS:
Overall Officials: Corey A Siegel, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (14):
- United States (14):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - University of Maryland Medical Center, Baltimore, Maryland
  - Brigham and Women's Hospital, Chestnut Hill, Massachusetts
  - Minnesota Gastroenterology, Plymouth, Minnesota
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Long Island Clinical Research Associates, LLP, Great Neck, New York
  - Winthrop University Hospital, Mineola, New York
  - Mount Sinai Medical Center, New York, New York
  - Charlotte Gastroenterology and Hepatology, PLLC, Charlotte, North Carolina
  - Ohio GI and Liver Institute, Cincinnati, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Zisman-Ilani Y, Thompson KD, Siegel LS, Mackenzie T, Crate DJ, Korzenik JR, Melmed GY, Kozuch P, Sands BE, Rubin DT, Regueiro MD, Cross R, Wolf DC, Hanson JS, Schwartz RM, Vrabie R, Kreines MD, Scherer T, Dubinsky MC, Siegel CA. Crohn's disease shared decision making intervention leads to more patients choosing combination therapy: a cluster randomised controlled trial. Aliment Pharmacol Ther. 2023 Jan;57(2):205-214. doi: 10.1111/apt.17286. Epub 2022 Nov 14. PMID 36377259